CLINICAL TRIAL: NCT00976352
Title: Phase I/II Trial of Diaphragm Delivery of Recombinant Adeno-Associated Virus Acid Alpha-Glucosidase (rAAV1-CMV-GAA) Gene Vector in Patients With Pompe Disease
Brief Title: Safety Study of Recombinant Adeno-Associated Virus Acid Alpha-Glucosidase to Treat Pompe Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PGTC PD-AAV004-N; P01HL059412-06 (NIH)
Record Dates: First submitted 2009-07-13; First posted 2009-09-14 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Pompe Disease
Keywords: Gene Therapy; Pompe Disease; Glycogen Storage Disease
MeSH Terms: conditions — Glycogen Storage Disease Type II; Glycogen Storage Disease | interventions — Pharmaceutical Preparations; Organization and Administration; Genetic Engineering

STUDY DESIGN:
Masking Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rAAV1-CMV-GAA administration-cohort 1 (Experimental): rAAV1-CMV-GAA (study agent) Administration: 1.0 x 10e12 vector genomes. The following study assessments/interventions will be completed: Respiratory Muscle Strength Training (RMST), Safety labs, pulmonary function testing.
  Interventions: Drug: rAAV1-CMV-GAA (study agent) Administration; Other: RMST
- rAAV1-CMV-GAA administration-cohort 2 (Experimental): rAAV1-CMV-GAA (study agent) Administration: 5.0 x 10e12 vector genomes Cohort 2 = 6 subjects. The following study assessments/interventions will be completed: Respiratory Muscle Strength Training (RMST), Safety labs, pulmonary function testing.
  Interventions: Drug: rAAV1-CMV-GAA (study agent) Administration; Other: RMST

INTERVENTIONS:
Drug: rAAV1-CMV-GAA (study agent) Administration — rAAV1-CMV-GAA via intramuscular injection into the diaphragm. Dose selection for cohort 1: 1.0 x 10e12 vector genomes Cohort 1 will have a total of 3 participants enrolled. Dose selection for cohort 2 and 3: 5.0 x 10e12 vector genomes rAAV1-CMV-GAA. Cohort 2 = 6 subjects.
  Other Names: Gene transfer; study agent (rAAV1-CMV-GAA)
Other: RMST — After enrollment and screening visit, the subject will be given a RMST prescription and will complete RMST for a minimum of 4 weeks prior to study agent administration. RMST prescription will be adjusted as needed at Day 14, 90, 180, and 270.
  Other Names: Respiratory Muscle Strength Training

SUMMARY:
Pompe disease is an inherited condition of acid alpha-glucosidase (GAA) deficiency resulting in lysosomal accumulation of glycogen in all tissues. Glycogen accumulation leads to muscle dysfunction and profound muscle weakness. A wide spectrum of disease is characteristic and the most severe patients have cardiorespiratory failure, often fatal in the first two years of life. Researchers have developed a way to introduce the normal GAA gene into muscle cells with the expectation that the GAA protein will be produced at levels sufficient to reduce glycogen accumulation. This study will evaluate the safety of the experimental gene transfer procedure in individuals with GAA deficiency. The study will also determine what dose may be required to achieve improvement in measures of respiratory function.

DETAILED DESCRIPTION:
The goal of the current study is to evaluate an experimental gene transfer procedure in which normal copies of the GAA gene are inserted into cells. In this study, a modified virus, adeno-associated virus (AAV), has been engineered to carry a normal copy of the GAA gene, known as rAAV1-CMV-hGAA, which is used to place normal copies of the GAA gene into diaphragm muscle cells. The purpose of this study is to evaluate the safety of rAAV1-CMV-hGAA delivery into individuals with GAA deficiency (Pompe Disease).

Participants currently using enzyme replacement therapy will continue to receive their regular medical regimen during the 12 month duration of the study. Participants will first attend a screening study visit to confirm study eligibility. Participants will then attend a 3-5 day inpatient visit, during which they will receive a series of intradiaphragmatic injections consisting of the study agent (rAAV1-CMV-hGAA). Follow-up study visits will occur on Days 14, 90, 180, 270 and 365. Participants will have yearly follow-up evaluations by either telephone or mail for a total of 15 years, or as required by the FDA and other regulatory agencies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 2-18 years of age.
* Have a diagnosis of Pompe, as defined by protein assay, DNA sequence of the acid alpha-glucosidase gene and clinical symptoms of the disease.
* Using assisted ventilation at baseline. Mechanical Ventilation is defined as any use of ventilation support, (including but not limited to BiPAP, CPAP), a minimum of 1 hours per day.
* Willing to discontinue aspirin, aspirin-containing products and other drugs that may alter platelet function, 7 days prior to dosing, resuming 24 hours after the dose has been administered.

Exclusion Criteria:

The subject must not:

* Have required acute, as distinguished from long-term, maintenance or chronic suppressive, oral or intravenous antibiotic therapy for a respiratory infection within 15 days prior to baseline screening.
* Have required oral or systemic corticosteroids within the last 15 days prior to baseline screening.
* Have a platelet count less than 75,000/ cu mm.
* Have an INR greater than 1.3.
* Serological evidence of hepatitis B, hepatitis C, or HIV positive.
* Be currently or within the past 30 days participating in any other research protocol involving investigational agents or therapies.
* Have received gene transfer agents within the past 6 months.
* Have history of platelet dysfunction, evidence of abnormal platelet function at screening or history of recent use of drugs that may alter platelet function which the subject is unable/unwilling to discontinue for study agent administration.
* Have any other concurrent condition which, in the opinion of the investigator, would make the subject unsuitable for the study.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry J Byrne, MD, PhD, Principal Investigator — University of Florida; Shelley Collins, MD, Principal Investigator — University of Florida
Locations (1):
- Shands at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fraites TJ Jr, Schleissing MR, Shanely RA, Walter GA, Cloutier DA, Zolotukhin I, Pauly DF, Raben N, Plotz PH, Powers SK, Kessler PD, Byrne BJ. Correction of the enzymatic and functional deficits in a model of Pompe disease using adeno-associated virus vectors. Mol Ther. 2002 May;5(5 Pt 1):571-8. doi: 10.1006/mthe.2002.0580. PMID 11991748
- [Background] Mah C, Cresawn KO, Fraites TJ Jr, Pacak CA, Lewis MA, Zolotukhin I, Byrne BJ. Sustained correction of glycogen storage disease type II using adeno-associated virus serotype 1 vectors. Gene Ther. 2005 Sep;12(18):1405-9. doi: 10.1038/sj.gt.3302550. PMID 15920463
- [Background] Mah C, Pacak CA, Cresawn KO, Deruisseau LR, Germain S, Lewis MA, Cloutier DA, Fuller DD, Byrne BJ. Physiological correction of Pompe disease by systemic delivery of adeno-associated virus serotype 1 vectors. Mol Ther. 2007 Mar;15(3):501-7. doi: 10.1038/sj.mt.6300100. Epub 2007 Jan 23. PMID 17245350
- [Background] Pauly DF, Fraites TJ, Toma C, Bayes HS, Huie ML, Hirschhorn R, Plotz PH, Raben N, Kessler PD, Byrne BJ. Intercellular transfer of the virally derived precursor form of acid alpha-glucosidase corrects the enzyme deficiency in inherited cardioskeletal myopathy Pompe disease. Hum Gene Ther. 2001 Mar 20;12(5):527-38. doi: 10.1089/104303401300042447. PMID 11268285
- [Background] Conlon TJ, Erger K, Porvasnik S, Cossette T, Roberts C, Combee L, Islam S, Kelley J, Cloutier D, Clement N, Abernathy CR, Byrne BJ. Preclinical toxicology and biodistribution studies of recombinant adeno-associated virus 1 human acid alpha-glucosidase. Hum Gene Ther Clin Dev. 2013 Sep;24(3):127-33. doi: 10.1089/humc.2013.147. PMID 24021025
- [Background] Byrne BJ. Pathway for approval of a gene therapy orphan product: treading new ground. Mol Ther. 2013 Aug;21(8):1465-6. doi: 10.1038/mt.2013.157. No abstract available. PMID 23903569
- [Background] Corti M, Elder M, Falk D, Lawson L, Smith B, Nayak S, Conlon T, Clement N, Erger K, Lavassani E, Green M, Doerfler P, Herzog R, Byrne B. B-Cell Depletion is Protective Against Anti-AAV Capsid Immune Response: A Human Subject Case Study. Mol Ther Methods Clin Dev. 2014;1:14033-. doi: 10.1038/mtm.2014.33. PMID 25541616
- [Result] Smith BK, Collins SW, Conlon TJ, Mah CS, Lawson LA, Martin AD, Fuller DD, Cleaver BD, Clement N, Phillips D, Islam S, Dobjia N, Byrne BJ. Phase I/II trial of adeno-associated virus-mediated alpha-glucosidase gene therapy to the diaphragm for chronic respiratory failure in Pompe disease: initial safety and ventilatory outcomes. Hum Gene Ther. 2013 Jun;24(6):630-40. doi: 10.1089/hum.2012.250. PMID 23570273
- [Derived] Byrne BJ, Falk DJ, Clement N, Mah CS. Gene therapy approaches for lysosomal storage disease: next-generation treatment. Hum Gene Ther. 2012 Aug;23(8):808-15. doi: 10.1089/hum.2012.140. PMID 22794786

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Pediatric Neuromuscular Disorders Clinic at the University of Florida. Subjects were also self-referred from the ClinicalTrials.gov listing.
Pre-assignment Details: All subjects underwent a screening process for eligibility determination as well as for safety evaluations.
Period: Overall Study
Arm/Group | rAAV1-CMV-GAA Administration-cohort 1 | rAAV1-CMV-GAA Administration-cohort 2
Started | 3 | 10
Completed | 3 | 6 (Last evaluation of last subject in cohort.)
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rAAV1-CMV-GAA Administration-cohort 1 | rAAV1-CMV-GAA Administration-cohort 2 | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 6 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: months] | 90 [66 to 108] | 67.3 [30 to 180] | 74.8 [30 to 180]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessments of the rAAV1-CMV-GAA (Study Agent), Changes Post Study Agent Administration.
Description: Change in Adeno-associated virus (AAV) antibody level; Change in Alglucosidase alpha (GAA) Antibody level
Time Frame: Change from baseline to 365 post study agent administration.
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | rAAV1-CMV-GAA Administration-cohort 1 | rAAV1-CMV-GAA Administration-cohort 2
Number analyzed (Participants) | 3 | 6
mU/mL
  AAV1antibody Level -Screening | 40,031 (65324.18978) | 29,638 (12395.02473)
  AAV1antibody Level - Day 365 | 5,509,882 (3051265.999) | 1,907,161 (3,189,557)
  GAA Antibody level - Screening | 415.6666667 (61.71169527) | 330.4 (271.1112318)
  GAA Antibody level - Day 365 | 504.3333333 (63.88531391) | 494.3333333 (371.6481311)

2. Secondary Outcome: Maximal Inspiratory Pressure
Description: Median (range) Maximal Inspiratory Pressure (MIP), in cm H2O
Time Frame: Baseline and 365 post study agent administration
Measure: Median (Full Range); unit: cm H2O
Arm/Group | rAAV1-CMV-GAA Administration-cohort 1 | rAAV1-CMV-GAA Administration-cohort 2
Number analyzed (Participants) | 3 | 6
cm H2O
  Baseline | 6 [2 to 22] | 61 [3 to 85]
  Day 365 | 6 [2 to 19] | 56 [3 to 75]

3. Secondary Outcome: Evaluation of Ventilatory Performance Benefit of rAAV1-CMV-GAA Gene Transfer and Respiratory Muscle Strength Training (RMST) Compared to RMST Alone.
Description: Median (range) maximal inspiratory pressure, in cm H2O. Timeframe for RMST training was 90 days prior to rAAV1-CMV-GAA gene transfer. Timeframe for following subjects after rAAV1-CMV-GAA gene transfer was 365 days.
Time Frame: Screening, Baseline, and 365 post study agent administration.
Measure: Median (Full Range); unit: cm H2O
Groups:
- rAAV1-CMV-GAA Administration-cohort 1: rAAV1-CMV-GAA (study agent) Administration: 1.0 x 10e12 vector genomes. The following study assessments/interventions will be completed: Respiratory Muscle Strength Training (RMST), Safety labs, pulmonary function testing.
  rAAV1-CMV-GAA (study agent) Administration: rAAV1-CMV-GAA via intramuscular injection into the diaphragm. Dose selection for cohort 1: 1.0 x 10e12 vector genomes Cohort 1 will have a total of 3 participants enrolled. Dose selection for cohort 2 and 3: 5.0 x 10e12 vector genomes rAAV1-CMV-GAA. Cohort 2 = 6 subjects.
  RMST: After enrollment and screening visit, the subject will be given a RMST prescription and will complete RMST for a minimum of 4 weeks prior to study agent administration. RMST prescription will be adjusted as needed at Day 14, 90, 180, and 270 after dosing.
- rAAV1-CMV-GAA Administration-cohort 2: rAAV1-CMV-GAA (study agent) Administration: 5.0 x 10e12 vector genomes Cohort 2 = 6 subjects. The following study assessments/interventions will be completed: Respiratory Muscle Strength Training (RMST), Safety labs, pulmonary function testing.
  rAAV1-CMV-GAA (study agent) Administration: rAAV1-CMV-GAA via intramuscular injection into the diaphragm. Dose selection for cohort 1: 1.0 x 10e12 vector genomes Cohort 1 will have a total of 3 participants enrolled. Dose selection for cohort 2 and 3: 5.0 x 10e12 vector genomes rAAV1-CMV-GAA. Cohort 2 = 6 subjects.
  RMST: After enrollment and screening visit, the subject will be given a RMST prescription and will complete RMST for a minimum of 4 weeks prior to study agent administration. RMST prescription will be adjusted as needed at Day 14, 90, 180, and 270 after dosing.
Arm/Group | rAAV1-CMV-GAA Administration-cohort 1 | rAAV1-CMV-GAA Administration-cohort 2
Number analyzed (Participants) | 3 | 6
cm H2O
  Screening | 6.85 [1.6 to 26.1] | 60.8 [1.9 to 82.6]
  Baseline | 5.85 [1.55 to 22.85] | 60.8 [2.65 to 84.85]
  Day 365 | 5.7 [1.65 to 19.1] | 55.6 [2.9 to 75.1]

4. Secondary Outcome: Evaluation of Tidal Volume Benefit of rAAV1-CMV-GAA Gene Transfer and Respiratory Muscle Strength Training, Compared to Respiratory Muscle Strength Training Alone.
Description: Best effort tidal volume, referenced to body mass, without use of ventilator assistance. Timeframe for respiratory muscle strength training alone was 90 days prior to dosing, timeframe post adminstration of rAAV1-CMV-GAA was 365 days.
Time Frame: Screening, Baseline, and Day 365 post study agent administration
Measure: Median (Full Range); unit: mL/kg
Groups:
- rAAV1-CMV-GAA Administration-cohort 1; rAAV1-CMV-GAA Administration-cohort 2: RMST: After enrollment and screening visit, the subject will be given a RMST prescription and will complete RMST for a minimum of 4 weeks prior to study agent administration. RMST prescription will be adjusted as needed at Day 14, 90, 180, and 270 after dosing.
Arm/Group | rAAV1-CMV-GAA Administration-cohort 1 | rAAV1-CMV-GAA Administration-cohort 2
Number analyzed (Participants) | 3 | 6
mL/kg
  Screening | 2.8 [0.7 to 4.0] | 7.9 [.14 to 8.7]
  Baseline | 2.0 [0.4 to 4.1] | 7.3 [.16 to 11.7]
  Day 365 | 3.4 [.71 to 4.3] | 9.1 [.18 to 13.3]

ADVERSE EVENTS:
Time Frame: Data on adverse events were collected on all subjects for 1 year after dosing.
Arm/Group | rAAV1-CMV-GAA Administration-cohort 1 | rAAV1-CMV-GAA Administration-cohort 2
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/9
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAAV1-CMV-GAA Administration-cohort 1 (N=3) | rAAV1-CMV-GAA Administration-cohort 2 (N=9)
Right-sided spontaneous pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bilateral pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bilateral pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Right upper lobe collapse with respiratory distress and Clostridium difficile gastritis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) — The subject was hospitalized 10 months post-dosing during the first occurrence of this SAE. The same subject was hospitalized 11 months post-dosing for an acute episode of desaturation, right upper lobe collapse, recurrent gastritis.
Bacteremia accompanied by fever (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Occurred 3 months post dosing. This unexpected event was determined to be unrelated to the test article and study procedures.
Desaturation Episode (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hospitalization: dehydration, increased work of breathing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hospitalization: dehydration, increased work of breathing
Hospitalization (General disorders) | 0 (0) | 3 (3)
hospitalization, worsening CHF, pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — hospitalization, worsening CHF, pulmonary edema
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAAV1-CMV-GAA Administration-cohort 1 (N=3) | rAAV1-CMV-GAA Administration-cohort 2 (N=9)
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Pneumothorax/Capnothorax (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 3 (3)
respiratory symthomps (Respiratory, thoracic and mediastinal disorders) | 3 (10) | 7 (18) — Cough, Increased secretions, cold symptoms, desaturation, oxygen requirement,Increased work of breathing, wheezing and Diminished breath sounds
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
fever, bacteremia, Dehydration (General disorders) | 3 (4) | 5 (7) — fever, bacteremia, Dehydration
Pulmonary and chest problems (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) — lung contusion, chest problems,
Reflux and Diarrhea, G-tube problems (Gastrointestinal disorders) | 3 (3) | 4 (8) — change to bowel and bladder regimen, Reflux and Diarrhea, stomach virus, G-tube problems, Abdominal abscess
Pain (General disorders) | 2 (3) | 4 (9) — pain, cramps
Skin issue (Skin and subcutaneous tissue disorders) | 2 (5) | 3 (6) — Swelling, rash,
Trachestomy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ear infection and fluids (Ear and labyrinth disorders) | 1 (2) | 2 (2)
eye infection (Eye disorders) | 0 (0) | 1 (2) — chalazion
Contracturs and scoliosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (3)
Hypokalemia and Hypoglycemia (General disorders) | 1 (1) | 1 (2)
Tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
urinary issues (Renal and urinary disorders) | 1 (1) | 2 (2) — Increased difficulty urinating, positional; infections
Nosebleed (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes